CLINICAL TRIAL: NCT02090868
Title: How the Introduction of an Oral Intake Screening Tool Can Benefit Patients Receiving Non-Invasive Ventilation
Brief Title: An Oral Intake Screening Tool for Patients Receiving Non-Invasive Ventilation
Status: Withdrawn | Type: Observational
Why Stopped: No patients recruited due to decreased levels of patients requiring non-invasive ventilation during the study.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 13IC0065
Record Dates: First submitted 2013-05-02; First posted 2014-03-18 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Patients Requiring Non-invasive Ventilation
Keywords: Non-Invasive Ventilation; Bi-Level Positive Airway Pressure; Continuous Positive Airway Pressure; Critical Care; Nutrition; Malnutrition; Staff attitudes, knowledge and beliefs
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre Introduction: Pre tool introduction cohort 22 patient participants who will receive standard care (no patients were recruited)
- Nurses: 12 nurse participants who will take part in 2 focus group interviews and a teaching session (6 nurse participants were recruited)
- Post Introduction: Pre tool introduction cohort 22 patient participants who's ability to eat and drink orally will be assessed using the Oral Intake Screening Tool (no patient participants were recruited)
  Interventions: Other: Oral Intake Screening Tool

INTERVENTIONS:
Other: Oral Intake Screening Tool — A screening tool developed from a literature review and expert opinion. It will be used by nurses to assess patients receiving non-invasive ventilation ability to eat and drink orally and suggest what actions should be taken if they are unable to do so
  Groups: Post Introduction

SUMMARY:
This study aims to explore how the introduction of an oral intake screening tool can benefit patients requiring noninvasive ventilation. The Quality Care Commission has identified nutritional problems in hospital and there is much literature on the importance of nutrition when critically ill. Literature is short however concerning the specialized population of those requiring noninvasive ventilation and they are a high risk group of suffering from malnutrition.

This study will potentially benefit patients by improving their nutritional care through guided assessment and nurse training.

The study will use mixed methodology, a prospective cohort study and qualitative interviews. The prospective cohort study will collect data from patients prior to the tool introduction, the control group, and post the tool introduction, the exposure group. This will enable comparisons to be made between the exposure and the control groups.

Nurses will be interviewed in semi structured focus groups prior to tool introduction and post to identify themes and sub themes to give a deeper understanding of nutrition in hospital and to examine the use of the tool in practice.

Patients will be eligible if they are over 18 and requiring noninvasive ventilation and nurses will be eligible if they work on the high dependency unit. Patients will be visited daily and have four mid arm circumference measurements at day 1, day 3, day 7 and day 14. The other daily visits will involve collecting data, which is recorded as part of routine care.

Nurses will undergo 2 focus group interviews and a teaching session. The study will take place at St Mary's hospital funded by Imperial College London. The study will be split into two periods with a two week gap in between. Each period will last until 22 patient participants have been recruited.

DETAILED DESCRIPTION:
No patients were recruited to the study due to decreased levels of patients requiring non-invasive ventilation during the study period and time constraints owing to an academic award submission date. Six nurse participants were recruited to the study and underwent two focus group interviews, one prior to tool implementation and one post.

ELIGIBILITY:
Patients

Inclusion Criteria:

* over 18 years old
* require non-invasive ventilation as defined by the protocol

Exclusion Criteria:

* Patients on the Liverpool Care Pathway
* Patients requiring nocturnal non-invasive ventilation only
* Patients with a tracheostomy
* Patients with a nasogastric feeding tube insitu on admission
* Patients with a PEG/RIG tube insitu on admission

Staff

Inclusion Criteria:

* full time employees
* work in the medical high dependency unit

Exclusion Criteria:

* staff only working bank or agency shifts on the medical high dependency unit
* staff who have not had formal high dependency/critical care training
* staff who do not work more than 5 shifts per month in the medical high dependency unit
* staff who have not held a full time post on Douglas Acute Admissions Unit for more than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients; Medical High Dependency Unit Patients Staff; Full time employees on the Douglas Acute Admission Unit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mid Arm Circumference Change | Day 1, 3, 7, 14

SECONDARY OUTCOMES:
Fluid Intake Change | Daily over 14 days
  fluid intake from all sources eg intravenous, nasogastric, oral
fluid balance change | daily for 14 days
  fluid intake minus fluid output
New formation of or worsening of existing pressure sores | daily for 14 days
new diagnosis of aspiration pneumonia | daily for 14 days
number of days requiring non-invasive ventilation | 14 days
number of days requiring level 2 care | 14 days
length of hospital stay | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - St Marys Hospital, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No